CLINICAL TRIAL: NCT04228120
Title: The Effects of a Self-regulation Program on Self-care Behaviour in Patients With Heart Failure: A Randomized Controlled Trial
Brief Title: Effects of a Self-regulation Program on Self-care Behaviour of Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Ai-Fu Chiou, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CGH-P103008
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
Keywords: Self-care behaviour; Self-regulation; Heart Failure
MeSH Terms: conditions — Heart Failure; Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The programme consisted of one 20-to-30-minute, face-to-face individual education session related to self-regulation and problem-solving processes that was performed in accordance with the patient's plan. Furthermore, eight 15- to 20-minute telephone follow-up counselling sessions were delivered twice per week for four weeks.
  Interventions: Behavioral: self-regulation programme
- control group (No Intervention): routine care

INTERVENTIONS:
Behavioral: self-regulation programme — The programme consisted of one 20-to-30-minute, face-to-face individual education session related to self-regulation and problem-solving processes that was performed in accordance with the patient's plan. Furthermore, eight 15- to 20-minute telephone follow-up counselling sessions were delivered twice per week for four weeks.
  Arms: intervention group

SUMMARY:
This RCT study aims to examine the effects of a self-regulation programme on the self-care behaviour and quality of life of patients with heart failure. The following hypothesis was tested: Heart failure patients who receive the self-regulation program will report significant improvements in self-care behaviours after four weeks of the self-regulation programme. In contrast, patients in the control group showed no significant differences.

DETAILED DESCRIPTION:
Eight two patients with heart failure were randomly assigned into the intervention (n = 41) or control group (n = 41). The intervention group participated in a 4-week self-regulation programme, including 20 to 30 minutes of individual self-regulation education and 15 to 20 minutes of telephone follow-up twice per week for four weeks. The control group received only routine outpatient care. Self-care behaviour was measured by the Self-Care of Heart Failure Index at baseline, 4 weeks and 8 weeks after patients were enrolled. Quality of life was measure with the Minnesota Living with Heart Failure questionnaire

ELIGIBILITY:
Inclusion Criteria:

* aged 20 years or older with heart failure diagnosed by a cardiologist (ICD-9:428)
* willing to communicate and participate in this study
* had clear consciousness

Exclusion Criteria:

* a diagnosis of cancer
* a diagnosis of mental illness including anxiety and depression
* had cognitive impairment
* a diagnosis of lung disease, such as asthma or chronic obstructive pulmonary disease
* a diagnosis of renal failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in three self-care behaviour subscale scores | 4 weeks and 8 weeks
  Changes from baseline Self-Care of Heart Failure Index (version 6.2) with three subscales: self-care maintenance, self-care management, and self-care confidence, at 4 weeks and 8 weeks. Each subscale score ranges from 0 to 100, with higher scores indicating better self-care behaviour.

SECONDARY OUTCOMES:
Change in quality of life scores | 4 weeks and 8 weeks
  Change from baseline Minnesota Living with Heart failure questionnaire scores at 4 weeks and 8 weeks. The total score range is 0-105; a higher score indicates lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ai-Fu Chiou, Ph.D, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: No